CLINICAL TRIAL: NCT00250939
Title: Single-center, Open-label Study of Safety, Pharmacokinetics and Efficacy of rhGAA in Patients With Late-Onset Pompe Disease
Brief Title: A Study of rhGAA in Patients With Late-Onset Pompe Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU02804
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Pompe Disease (Late-onset); Glycogen Storage Disease Type II (GSD-II); Acid Maltase Deficiency Disease; Glycogenosis 2
Keywords: Glycogen Storage Disease Type II; GSD-II; Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Myozyme

INTERVENTIONS:
Biological: Myozyme — 20 mg/kg qow
  Other Names: alglucosidase alfa

SUMMARY:
Pompe disease (also known as glycogen storage disease Type II) is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. The overall objective is to evaluate the safety, pharmacokinetics (PK) and efficacy of Myozyme treatment.

ELIGIBILITY:
Inclusion Criteria:

* patient's legally authorized guardian(s) must provide signed, informed consent prior to performing any study-related procedures; patient's signature required if patient understands informed consent
* patient must have a diagnosis of Pompe disease based on deficient endogenous GAA activity or GAA gene mutations
* patient must have demonstrable muscle weakness
* patient must be greater than or equal to five years of age and younger than eighteen years of age
* patient must be able to provide 3 reproducible FVC tests in sitting position during screening
* patient must perform muscle function testing
* patient must ambulate 10 meters (assistive devices permitted)
* patient and legal guardian must comply with the clinical protocol

Exclusion Criteria:

* patient requires the use of invasive ventilatory support
* patient requires the use of noninvasive ventilatory support while awake and in an upright position
* patient has received enzyme replacement therapy with GAA from any source
* patient has used an investigational product within 30 days prior to study enrollment, or is currently enrolled in another clinical or observational study
* patient has a medical condition, serious intercurrent illness, or other extenuating circumstance that, may significantly interfere with study compliance, including all prescribed evaluations and follow-up activities
* Female patients pregnant, lactating or unwilling to practice birth control methods during study
* Male patients unwilling to use barrier contraceptives during study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2005-02; Primary Completion 2006-07 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
safety and PK profile rhGAA | 74 weeks
FVC | 74 weeks
MMT | 74 weeks
Effect of treatment on muscle function | 74 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Sophia Kinderziekenhuis, Erasmus MC, Rotterdam, Netherlands